CLINICAL TRIAL: NCT01710527
Title: AN OPEN LABEL, BALANCED, RANDOMIZED, TWO-TREATMENT, TWO-PERIOD, TWO-SEQUENCE, CROSSOVER, SINGLE ORAL DOSE, BIOEQUIVALENCE STUDY OF METFORMIN 500 MG TABLETS MANUFACTURED BY SAVIPHARM J.S.C, VIETNAM AND GLUCOPHAGE® 500 MG TABLETS MANUFACTURED BY MERCK SANTE S.A.S.2, RUE DU PRESSOIR VERT-45400 SEMOY-FRANCE AND BE REGISTERED IN VIETNAM IN HEALTHY, ADULT, HUMAN MALE SUBJECTS UNDER FASTING CONDITION
Brief Title: BE Study of Metformin GSK 500mg
Acronym: BA/BE 173/11
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 116723
Record Dates: First submitted 2012-09-27; First posted 2012-10-19 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-04

CONDITIONS: Diabetic Foot
Keywords: Healthy Volunteers
MeSH Terms: conditions — Diabetic Foot | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin 500mg (Other): Cross over, two treatment, two period, two sequence, cross over, single dose
  Interventions: Drug: Metformin 500mg; Drug: Glucophage 500mg
- Glucophage 500mg (Other): Cross over, two treatment, two period, two sequence, sigle dose
  Interventions: Drug: Metformin 500mg; Drug: Glucophage 500mg

INTERVENTIONS:
Drug: Metformin 500mg — EVALUATE BIOEQUIVALENCE BETWEEN METFORMIN 500 MG TABLETS MANUFACTURED BY SAVIPHARM J.S.C, VIETNAM AND GLUCOPHAGE® 500 MG TABLETS MANUFACTURED BY MERCK SANTE S.A.S.2, RUE DU PRESSOIR VERT-45400 SEMOY-FRANCE AND BE REGISTERED IN VIETNAM IN HEALTHY, ADULT, HUMAN MALE SUBJECTS UNDER FASTING CONDITION
Drug: Glucophage 500mg — EVALUATE BIOEQUIVALENCE BETWEEN METFORMIN 500 MG TABLETS MANUFACTURED BY SAVIPHARM J.S.C, VIETNAM AND GLUCOPHAGE® 500 MG TABLETS MANUFACTURED BY MERCK SANTE S.A.S.2, RUE DU PRESSOIR VERT-45400 SEMOY-FRANCE AND BE REGISTERED IN VIETNAM IN HEALTHY, ADULT, HUMAN MALE SUBJECTS UNDER FASTING CONDITION

SUMMARY:
A randomized, balanced, open label, crossover, two period, two treatment, two sequence, single dose, oral bioequivalence study under fasting condition. It is a pivotal study.

To demonstrate the bioequivalence of Metformin 500 mg tablets manufactured by Savipharm J.S.C, Vietnam and Glucophage® 500 mg tablets of MERCK SANTE in healthy adult human male subjects under fasting condition and to monitor the safety of the study subjects.

DETAILED DESCRIPTION:
Sample Size Estimation Assuming the formulation ratio (T/R) 95-105% and with the maximum observable intra subject variability for Metformin is 22% (based on literature), a sample size of 29 subjects would be sufficient to prove bioequivalence between the two formulations with power of at least 90%. Hence, total 32 subjects will be enrolled in the study considering withdrawal and dropouts.

Hence, 32 healthy adult human male subjects will be enrolled. Adverse Events The investigator or site staff is responsible for detecting, documenting and reporting events that meet the definition of an AE or SAE.

AEs will be collected from the start of Study Treatment and until the follow-up contact. Medical occurrences that begin prior to the start of study treatment but after obtaining informed consent may be recorded on the Medical History/Current Medical Conditions CRF.

SAEs will be collected over the same time period as stated above for AEs. However, any SAEs assessed as related to study participation (e.g. study treatment, protocol-mandated procedures, invasive tests, or change in existing therapy) or related to a GSK concomitant medication will be recorded from the time a subject consents to participate in the study up to and including any follow-up contact. All SAEs will be recorded and reported to the sponsor within 24 hours.

Investigators are not obligated to actively seek AEs or SAEs in former study participants. However, if the investigator learns of any SAE, including a death, at any time after a subject has been discharged from the study, and he considers the event reasonably related to the study treatment or study participation, the investigator would promptly notify the sponsor.

All serious adverse events will be informed to the sponsor within 24 hrs and to the IEC within 7 working days. Any unexpected serious adverse event (SAE) occurring during a clinical trial should be communicated promptly (within 14 calendar days) by the Sponsor/CRO to the Licensing Authority.

Any follow-up information on a previously reported SAE will also be reported to the sponsor within 24 hours.

If the investigator does not have all information regarding an SAE, he/she will not wait to receive additional information before notifying the sponsor of the event and completing the appropriate data collection tool. The investigator will always provide an assessment of causality at the time of the initial report.

Screening procedures: Demographic data, medical and medication histories, complete physical examination, height, weight and BMI as well as 12 lead ECG, chest X-ray [PA view], vital signs [blood pressure, pulse rate, respiratory rate and oral temperature], hematology, biochemistry, HIV 1 & 2, Hepatitis B and C, RPR test for Syphilis and urine analysis will be done at screening.

Urine drug screen, Liver chemistry test and breath alcohol test to be done prior to each check-in.

Breath alcohol test to be done prior to each ambulatory visit blood collection. Liver chemistry test to be done at the end of each period. Housing: The study subjects will be housed at least 11 h prior to drug administration until after the 24 h blood sampling in each study period. The housing will be followed by one ambulatory visits [36.0 hr post dose] for each period.

Washout: At least 7 days, but not exceeding 14 days between two dosing days. Treatment arms: Test: A single dose of Metformin 500 mg tablet manufactured by Savipharm J.S.C, Vietnam.

Reference: A single dose of Glucophage® 500 mg tablet of Merck Sante, France Drug administration: As per the randomization schedule, one tablet of either test or reference product will be orally administered to each subject in each period in sitting posture, after an overnight fast of at least 10 h.

To avoid hypoglycemic episodes, the investigational products will be administered with 240 mL of a 20% glucose solution in water, followed by 60 mL of the glucose solution administered every 15 min for up to 4 h after dosing.

Subjects will be instructed not to chew or crush the tablet but should be swallowed. Compliance for dosing will be assessed by identification of subjects with subject ID card, identification of label on investigational product to confirm correct allocation of treatment and checking the oral cavity immediately after dosing.

Restrictions: Subjects will remain in upright position [sitting or ambulatory] for two hours after dosing in each period except when clinically indicated to change the posture. The subjects will fast for at least 10 h prior to dosing and 4 h post-dose. Water will be permitted ad libitum except for 1 h before and until 1 h after post dose. During 1 hr post dose water restriction a, 60 mL of 20% glucose solution will be administered every 15 min to the study subjects.

In each period of the study, 18 blood samples of 6 mL each will be collected in K2EDTA vacutainers via an indwelling catheter placed in one of the forearm veins. Heparin-lock technique will be used to prevent clotting of blood in the indwelling catheter. Before each in-house blood sample is drawn through catheter, 0.5 mL of blood will be discarded so as to purge the heparin containing blood sample in the catheter. Blood can also be collected by direct venipuncture in case of cannula blockage, during ambulatory visits or for any other practical reasons. The two pre-dose blood samples will be collected within a period of 1 h before the drug administration. The post-dose blood samples will be collected at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0 and 36.0 h. The 36.0 h post dose blood samples will be collected during ambulatory visits by direct venipuncture. Immediately after collection of blood, the sample will be kept in ice bath. After collecting the blood samples from all the subjects at each sampling time point, samples will be centrifuged at 4oC with 3500 rpm for 10 minutes. The plasma samples will be separated and stored in pre-labeled polypropylene tubes at -70 ± 10°C pending assay. The time interval between sample collection and the start of centrifugation should not exceed more than 45 minutes. The blood sample collection, processing and analysis will be done under sodium monochromatic light.

The total volume of blood drawn including the volume necessary for the laboratory tests, PK sample analysis and the volume of blood discarded before each in house blood draw will be about 250 mL per subject for the entire study.

Subjects monitoring: Brief physical examination and vital signs [blood pressure, pulse rate and oral temperature] will be carried out and recorded at each check-in and at check-out. Vital signs [blood pressure and pulse rate] will also be recorded before dosing of investigational products, between 2 - 3, 9 - 10 and 36.0 h post dose. Vital signs should be done in sitting position after rest of at least 5 minutes. Physical examination and measurement of vital signs can also be carried out at any time during the conduct of the study if the Investigator/Doctor feels it necessary. In case of abnormality in pre-dose vital signs, Investigator based on his medical judgement will take the decision whether to dose the subject or not. During vitals recording each subject will be asked about his well-being. Also subject well-being questionnaire will be performed at 1.0 and 5.0 h post dose.

Post-study Procedures: Safety evaluation [complete physical examination, vital signs, hematology [except blood grouping & Rh typing] and biochemistry] will be done at the end of the clinical part of the study. In case of any withdrawals during the study safety assessment will be done at the time of withdrawal. In case of dropouts subjects will be asked to visit the facility to undergo safety assessments.

Pharmacokinetic Parameters: Cmax, Tmax, AUC0-t, AUC0-∞, AUC%_Extrap, Kel and t1/2 Analytical Methods: Metformin in plasma will be estimated using validated LC-MS/MS method.

Statistical Methods: Statistical analyses will be done using SAS® version 9.2 or higher. Analysis of variance [ANOVA] for log-transformed pharmacokinetic parameters [Cmax, AUC0-t and AUC0-∞], two one-sided tests [Schuirmann] for bioequivalence, power, ratio and 90% confidence interval for log-transformed pharmacokinetic parameters - Cmax, AUC0-t and AUC0-∞ will be performed.

Standards for Bioequivalence: The calculated 90% Confidence Interval for the test to reference ratio of Metformin should fall within the range of 80%-125% for log transformed Cmax, AUC0-t and AUC0-∞ for the conclusion of bioequivalence.

ELIGIBILITY:
Inclusion Criteria

* Healthy adult male human subjects within the age range of 18 to 45 years inclusive.
* Weight not less than 50 kg.
* Normal BMI [18.5 to 24.99 kg/m2 inclusive].
* Willingness and capability to provide written informed consent to participate in the study.
* Free of significant diseases or clinically significant abnormal findings based on medical history, physical examination, laboratory evaluations, 12-lead ECG, Chest X-ray [PA view].
* Absence of disease markers of HIV 1 and 2, Hepatitis B and C and Syphilis.
* AST, ALT, alkaline phosphatase and bilirubin </=1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* ECG normal for morphology and measurements. QTcB or QTcF < 450 msec or QTc < 480 msec in subjects with Bundle Branch Block, based on an average from three ECGs obtained over a brief recording period.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed below. This criterion must be followed from the time of the first dose of study medication until one week of last dose administration.

  * Condom plus partner use of a highly effective contraceptive such as occlusive cap (diaphragm or cervical/vault cap) plus spermicidal agent (foam/gel/film/cream/suppository), oral contraceptive, injectable progesterone, implant of etonogestrel or levonorgestrel, estrogenic vaginal ring, percutaneous contraceptive patches, or intrauterine device.

OR

* Abstinence, defined as sexual inactivity consistent with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g. calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria

* History or presence of significant: Cardiovascular, pulmonary, hepatic, renal, hematological, gastro-intestinal, endocrine, immunologic, dermatologic, neurological, psychiatric disease.
* History or presence of significant:

  * Alcohol dependence, alcohol abuse during past one year.
  * Drug abuse [Marijuana [THC], Cocaine, Morphine, Benzodiazepines, Barbiturates and Amphetamine] for the last 6 months.
  * Smoking of more than 5 cigarettes per day or consumption of other forms of tobacco containing products.
  * Asthma, urticaria or other allergic type reactions after taking aspirin or any other drug.
  * Ulceration or history of gastric and / or duodenal ulcer.
  * Jaundice in the past 6 months.
* Bleeding disorder.
* Allergy to the test drug or any drug chemically similar to the drug or to the excipients of the products under investigation.
* Donation of 500 mL or more blood within 8 weeks prior to receiving the first dose of study drug.
* Subjects who have participated in another clinical study in the past 3 months prior to commencement of this study.
* Any difficulty in accessibility of forearm veins for cannulation or blood sampling.
* Refusal to abstain from food for at least 10 h prior to drug administration and for at least 4 h post dose in each period.
* Refusal to abstain from fluid for at least 1 h prior to and 1 h post each dose except 20 % glucose solution given after dosing.
* Positive breath alcohol test result found on the day of check-in.
* Positive urine test result for drug of abuse found on the day of check-in.
* History of difficulty in swallowing tablet.
* Use of any concomitant medication [including over-the-counter products, vitamins etc.] for 14 days preceding the study drug administration.
* Use of drugs which induce or inhibit metabolizing enzymes within 30 days prior to receiving the first dose of study medication.

Other Eligibility Criteria Considerations To assess any potential impact on subject eligibility with regard to safety, the investigator must refer to the product data sheet for detailed information regarding warnings, precautions, contraindications, adverse events, and other significant data pertaining to the product being used in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05-09 (Actual); Primary Completion 2012-05-18 (Actual); Study Completion 2012-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Background] GSK has concluded that it is not feasible to publish this study in a peer-reviewed scientific journal because the nature of the study is unlikely to be of interest to a journal. GSK is providing a results summary with a conclusion.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted on 32 adult healthy male participants, aged between 18 and 45 years, at a single site of India from 9 May 2012 to 18 May 2012. During each study period participants received test (treatment T-Metformin tablet) and reference (treatment R-Glucophage® tablet) products.
Pre-assignment Details: A total of 32 participants were randomized in the period I to receive test (treatment T-Metformin 500 milligram [mg] tablet) or reference (treatment R-Glucophage 500 mg tablet).
Groups:
- Treatment T-Metformin 500mg, Then Treatment R-Glucophage 500mg: Participants received one tablet of treatment T (Metformin 500 mg tablet) given with 250 mL of 20% glucose solution in water followed by 60 mL of the glucose solution administered every 15 minutes (min) for up to 4 hours after dosing according to a plan of randomization. After a washout period of 7 days, participants then received one tablet of treatment R (Glucophage 500 mg tablet) given with 240 mL of 20% glucose solution in water followed by 60 mL of the glucose solution administered every 15 min for up to 4 hours after dosing. Participants were admitted the night before study drug administration, supervised for at least 10 hours of overnight fasting, and confined until collecting 24 hour post-dose blood sample during study drug administration of each period. The study drug administration took place between 8:00 ante meridiem (am) and 8:30 am on Day 1 (dosing day) of each study period.
- Treatment R-Glucophage 500mg, Then Treatment T-Metformin 500mg: Participants received one tablet of treatment R (Glucophage 500 mg tablet) given with 250 mL of 20% glucose solution in water followed by 60 mL of the glucose solution administered every 15 min for up to 4 hours after dosing according to a plan of randomization. After a washout period of 7 days, participants then received one tablet of treatment T (Metformin 500 mg tablet) given with 240 mL of 20% glucose solution in water followed by 60 mL of the glucose solution administered every 15 min for up to 4 hours after dosing. Participants were admitted the night before study drug administration, supervised for at least 10 hours of overnight fasting, and confined until collecting 24 hour post-dose blood sample during study drug administration of each period. The study drug administration took place between 8:00 am and 8:30 am on Day 1 (dosing day) of each study period.
Period: Period 1: Intervention Period 1
Arm/Group | Treatment T-Metformin 500mg, Then Treatment R-Glucophage 500mg | Treatment R-Glucophage 500mg, Then Treatment T-Metformin 500mg
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0
Period: Period 2: Washout Period (7 Days)
Arm/Group | Treatment T-Metformin 500mg, Then Treatment R-Glucophage 500mg | Treatment R-Glucophage 500mg, Then Treatment T-Metformin 500mg
Started | 16 | 16
Completed | 16 | 15
Not Completed | 0 | 1
Not completed — Personal reasons | 0 | 1
Period: Period 3: Intervention Period 2
Arm/Group | Treatment T-Metformin 500mg, Then Treatment R-Glucophage 500mg | Treatment R-Glucophage 500mg, Then Treatment T-Metformin 500mg
Started | 16 | 15
Completed | 16 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment T-Metformin 500 mg + Treatment R-Glucophage 500 mg: In each period of the study, participants received one tablet of treatment T (Metformin 500 mg tablet) or treatment R (Glucophage 500 mg tablet), with 240 mL of 20% glucose solution in water followed by 60 mL of the glucose solution administered every 15 min for up to 4 hours after dosing according to a plan of randomization. Participants were admitted the night before study drug administration, supervised for at least 10 hours of overnight fasting, and confined until collecting 24 hour post-dose blood sample during study drug administration of each period. The study drug administration took place between 8:00 am and 8:30 am on Day 1 (dosing day) of each study period. The two treatment periods were separated by a washout period of 7 days.
Arm/Group | Treatment T-Metformin 500 mg + Treatment R-Glucophage 500 mg
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26.19 (4.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 32
Region of Enrollment [Number; unit: Participants]
  India | 32

OUTCOME MEASURES:

1. Primary Outcome: Mean Maximal Measured Plasma Concentration (Cmax) After a Single Dose
Description: Plasma samples for pharmacokinetic (PK) analysis were drawn at indicated time points of each treatment period. Cmax was defined as maximal measured plasma concentration over the time span specified.
Time Frame: Pre- dose (0.0 hour), post-dose at 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0 and 36.0 hour in each period.
Population: PK population was defined as all participants who had a PK measurement available. Data is presented for the participants available at the time of assessment.
Measure: Mean (Standard Deviation); unit: Nanogram per milliltre (ng/mL)
Groups:
- Treatment T-Metformin 500 mg: In each period of the study, participants received one tablet of treatment T (Metformin 500 mg tablet), with 240 mL of 20% glucose solution in water followed by 60 mL of the glucose solution administered every 15 min for up to 4 hours after dosing either in sequence of treatment T/R or treatment R/T according to a plan of randomization. Participants were admitted the night before study drug administration, supervised for at least 10 hours of overnight fasting, and confined until collecting 24 hour post-dose blood sample during study drug administration of each period. The study drug administration took place between 8:00 am and 8:30 am on Day 1 (dosing day) of each study period. The two treatment periods were separated by a washout period of 7 days.
- Treatment R- Glucophage 500 mg: In each period of the study, participants received one tablet of treatment R (Glucophage 500 mg tablet), with 240 mL of 20% glucose solution in water followed by 60 mL of the glucose solution administered every 15 min for up to 4 hours after dosing either in sequence of treatment T/R or treatment R/T according to a plan of randomization. Participants were admitted the night before study drug administration, supervised for at least 10 hours of overnight fasting, and confined until collecting 24 hour post-dose blood sample during study drug administration of each period. The study drug administration took place between 8:00 am and 8:30 am on Day 1 (dosing day) of each study period. The two treatment periods were separated by a washout period of 7 days.
Arm/Group | Treatment T-Metformin 500 mg | Treatment R- Glucophage 500 mg
Number analyzed (Participants) | 31 | 31
Nanogram per milliltre (ng/mL) | 962.728 (246.0751) | 985.257 (223.1331)
Statistical Analysis 1: Comparison: Treatment T-Metformin 500 mg vs Treatment R- Glucophage 500 mg; Test type: Non-Inferiority or Equivalence — Bioequivalence of Treatment T-Metformin 500 mg with Treatment R- Glucophage 500 mg was concluded if the 90% confidence intervals for the ratio of log transformed Cmax fell within the acceptance range of 80 to 125%; p = 0.3125, ANOVA; Ratio (%) = 96.85, 90% CI 2-sided [91.86 to 102.11] — Analysis was performed on log transformed geometric least square means

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUC0-t) and Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-infinity)
Description: Plasma samples for PK analysis were drawn at indicated time points of each treatment period.
  AUC0-t was calculated by the linear trapezoidal rule from measured data points from time of administration until the time of last quantifiable concentration. AUC0- infinity was estimated by linear trapezoidal rule and was sum of the AUC0-t and extrapolated to infinity by dividing the estimated last measurable plasma concentration by elimination rate constant. The AUC0- infinity was the sum of the estimated and extrapolated parts.
Time Frame: as for outcome 1
Population: PK population. Data is presented for the participants available at the time of assessment.
Measure: Mean (Standard Deviation); unit: ng*hour/mL
Arm/Group | Treatment T-Metformin 500 mg | Treatment R- Glucophage 500 mg
Number analyzed (Participants) | 31 | 31
ng*hour/mL
  AUC0-t | 7396.329 (1869.1737) | 7215.743 (1865.2930)
  AUC0-infinity | 7577.176 (1856.9193) | 7400.540 (1866.7596)
Statistical Analysis 1: Comparison: Treatment T-Metformin 500 mg vs Treatment R- Glucophage 500 mg; Comparison of Treatment T-Metformin 500 mg and Treatment R- Glucophage 500 mg for AUC0-t; Test type: Non-Inferiority or Equivalence — Bioequivalence of Treatment T-Metformin 500 mg with Treatment R- Glucophage 500 mg was concluded if the 90% confidence intervals for the ratio of log transformed AUC0-t fell within the acceptance range of 80 to 125%; p = 0.2701, ANOVA; Ratio (%) = 102.52, 90% CI 2-sided [98.74 to 106.45]
Statistical Analysis 2: Comparison: Treatment T-Metformin 500 mg vs Treatment R- Glucophage 500 mg; Comparison of Treatment T-Metformin 500 mg and Treatment R- Glucophage 500 mg for AUC0-infinity; Test type: Non-Inferiority or Equivalence — Bioequivalence of Treatment T-Metformin 500 mg with Treatment R- Glucophage 500 mg was concluded if the 90% confidence intervals for the ratio of log transformed AUC0-infinity fell within the acceptance range of 80 to 125%; p = 0.2702, ANOVA; Ratio (%) = 102.44, 90% CI 2-sided [98.78 to 106.23] — Analysis was performed on log transformed geometric least square means

3. Primary Outcome: Time of the Maximum Plasma Concentration (T-max) Over Period
Description: Plasma samples for PK analysis were drawn at indicated time points of each treatment period. If the maximum value occurs at more than one point T-max was defined as the first time point with this value.
Time Frame: as for outcome 1
Population: PK population. Data is presented for the participants available at the time of assessment.
Measure: Median (Standard Deviation); unit: hour
Arm/Group | Treatment T-Metformin 500 mg | Treatment R- Glucophage 500 mg
Number analyzed (Participants) | 31 | 31
hour | 3.00 (0.910) | 3.00 (0.991)

4. Primary Outcome: Terminal Half-life (T-half) Over Period
Description: Plasma samples for PK analysis were drawn at indicated time points of each treatment period. The elimination or terminal half-life was calculated by dividing 0.693 (natural logarithm of 2) with elimination rate constant obtained as semi logarithmic plot of the plasma concentration versus time.
Time Frame: as for outcome 1
Population: PK population. Data is presented for the participants available at the time of assessment.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Treatment T-Metformin 500 mg | Treatment R- Glucophage 500 mg
Number analyzed (Participants) | 31 | 31
hour | 3.84 (0.511) | 3.86 (0.549)

5. Primary Outcome: Percentage of Area Under Curve Extrapolated to Arrive at AUC0-infinity (AUC%_Extrapolated)
Description: Plasma samples for PK analysis were drawn at indicated time points of each treatment period. AUC%_Extrapolated was obtained by subtracting AUC0-t from AUC0-infinity divided by AUC0-infinity and multiplied by 100.
Time Frame: as for outcome 1
Population: PK population. Data is presented for the participants available at the time of assessment.
Measure: Mean (Standard Deviation); unit: Percentage of area
Arm/Group | Treatment T-Metformin 500 mg | Treatment R- Glucophage 500 mg
Number analyzed (Participants) | 31 | 31
Percentage of area | 2.604 (1.5408) | 2.684 (1.6589)

6. Primary Outcome: Apparent First-order Elimination or Terminal Rate Constant
Description: Plasma samples for PK analysis were drawn at indicated time points of each treatment period. The apparent first-order elimination or terminal rate constant was calculated from a semi logarithmic plot of the plasma concentration versus time. The parameter was calculated by linear least-square regression analysis using the last three (or more) non-zero plasma concentrations.
Time Frame: as for outcome 1
Population: PK population. Data is presented for the participants available at the time of assessment.
Measure: Mean (Standard Deviation); unit: 1/hour
Arm/Group | Treatment T-Metformin 500 mg | Treatment R- Glucophage 500 mg
Number analyzed (Participants) | 31 | 31
1/hour | 0.183 (0.0250) | 0.184 (0.0285)

7. Secondary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An AE is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or is a congenital anomaly/birth defect, may jeopardize the participant or may require medical or surgical intervention to prevent one of the other outcomes listed in this definition, associated with liver injury and impaired liver function defined as alanine aminotransferase >=3 x upper limit of normal (ULN), and total bilirubin >=2 x ULN or international normalized ratio >1.5.
Time Frame: Up to 38 days
Population: Safety population was defined as participants who received at least one dose of the study drug.
Measure: Number; unit: Participants
Arm/Group | Treatment T-Metformin 500 mg | Treatment R- Glucophage 500 mg
Number analyzed (Participants) | 32 | 32
Participants
  Any AE | 2 | 1
  Any SAE | 0 | 0

8. Secondary Outcome: Number of Participants With Abnormal Vital Sign Results
Description: Vital signs measurements (blood pressure, respiratory rate, pulse rate and oral temperature) were conducted during screening and during post study safety assessments. Vital signs measurement were also performed at each check-in and at checkout and were also recorded before dosing of study drug, between 2-3, 9-10 and 36.0 hour post-dose. Measurements were recorded in sitting position after rest of at least 5 min.
Time Frame: Up to 38 days
Population: Safety population.
Measure: Number; unit: Participants
Arm/Group | Treatment T-Metformin 500 mg | Treatment R- Glucophage 500 mg
Number analyzed (Participants) | 32 | 32
Participants | 0 | 0

9. Secondary Outcome: Number of Participants With Abnormal Periodic Physical Examination Results
Description: Brief physical examination was performed at each check-in, check-out and complete physical examination during screening and at the end of the clinical part of the study.
Time Frame: Up to 38 days
Population: Safety population.
Measure: Number; unit: Participants
Arm/Group | Treatment T-Metformin 500 mg | Treatment R- Glucophage 500 mg
Number analyzed (Participants) | 32 | 32
Participants | 0 | 0

10. Secondary Outcome: Assessment of Subject Well-being Questionnaire
Description: Subject well-being questionnaire was planned to be conducted at 1.0 and 5.0 hour post-dose. During vital sign recording each participants was planned to be asked about his well-being recorded during post study safety assessments. The data for this outcome measure was not collected during the study. Thus the results summary for this outcome measure was not produced.
Time Frame: Up to 38 days
Population: Safety population.
Arm/Group | Treatment T-Metformin 500 mg | Treatment R- Glucophage 500 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: AE's and SAE's were collected up to 38 days.
Description: Safety population was used.
Groups:
- Treatment T-Metformin 500 mg: In each period of the study, participants received one tablet of treatment T (Metformin 500 mg tablet), with 240 mL of 20% glucose solution in water followed by 60 mL of the glucose solution administered every 15 min for up to 4 h after dosing either in sequence of treatment T/R or treatment R/T according to a plan of randomization. Participants were admitted the night before study drug administration, supervised for at least 10 h of overnight fasting, and confined until collecting 24 h post-dose blood sample during study drug administration of each period. The study drug administration took place between 8:00 am and 8:30 am on Day 1 (dosing day) of each study period. The two treatment periods were separated by a washout period of 7 days.
- Treatment R- Glucophage 500 mg: In each period of the study, participants received one tablet of treatment R (Glucophage 500 mg tablet), with 240 mL of 20% glucose solution in water followed by 60 mL of the glucose solution administered every 15 min for up to 4 h after dosing either in sequence of treatment T/R or treatment R/T according to a plan of randomization. Participants were admitted the night before study drug administration, supervised for at least 10 h of overnight fasting, and confined until collecting 24 h post-dose blood sample during study drug administration of each period. The study drug administration took place between 8:00 am and 8:30 am on Day 1 (dosing day) of each study period. The two treatment periods were separated by a washout period of 7 days.
Arm/Group | Treatment T-Metformin 500 mg | Treatment R- Glucophage 500 mg
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 2/32 | 1/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment T-Metformin 500 mg (N=32) | Treatment R- Glucophage 500 mg (N=32)
Vomiting (Gastrointestinal disorders) | 1 | 0
Headache (General disorders) | 1 | 0
Tiredness (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.